CLINICAL TRIAL: NCT03745365
Title: A Comparative Study Between Sleeve Gastrectomy and Combined Sleeve Gastrectomy With Loop Bipartition (Short-term Outcomes).
Brief Title: Comparison Between Sleeve Gastrectomy and Loop Bipartition (Short-term Outcomes)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdou Gad Youssef, doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SG vs. SG with loop BP
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Loop Bipartition

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups according to the surgical procedure performed as follows:
  * Group A: Patients undergoing sleeve gastrectomy.
  * Group B: Patients undergoing combined sleeve gastrectomy with loop bipartition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sleeve gastrectomy (Experimental): The greater omentum is divided 5 cm from the pylorus with an energy device. The antral pouch is measured 2-6cm from the pylorus along greater curve as risk benefit ratio is best within these limits.
  Devascularization is continued up the greater curve of the stomach to the short gastric vessels with the help of the assistant who maintains traction and exposure during this process. Eventually, one reaches the left crus which is an important landmark of dissection. We selectively explore the hiatus of the symptomatic and endoscopically proven hiatus hernia , and the hernia should be reduced and repaired.
  Interventions: Procedure: loop bipartition
- sleeve gastrectomy with loop bipartition (Experimental): Sleeve gastrectomy is performed first, then a loop gastro-ileostomy 200-250 cm from doudeno-jejunal junction was created at the dependent part of the antrum with 2 layers of with stapler but without division of the 1st part of duodenum. The resultant stomach tube has two outlets, one to the first part of duodenum through the pylorus and one to the terminal ileum through the gastro-ileostomy. The staple line and anastomosis was tested with methylene blue. A drain is inserted.
  Interventions: Procedure: loop bipartition

INTERVENTIONS:
Procedure: loop bipartition — A loop gastro-ileostomy 250-300 cm from the ileocecal valve or 200-250 cm from duodeno-jejunal junction was created at the dependent part of the antrum with 2 layers of handsewn suture but without division of the 1st part of duodenum. The resultant stomach tube has two outlets, one to the first part of duodenum through the pylorus and one to the terminal ileum through the gastroileostomy.

SUMMARY:
Aim of the study is To compare short-term outcomes of sleeve gastrectomy operation with those of combined sleeve gastrectomy and loop bipartition procedure.

DETAILED DESCRIPTION:
Bariatric surgery has been shown to be the most effective and durable treatment for morbid obesity. Surgery results in significant weight loss and helps prevent, improve or resolve more than 40 obesity-related diseases or conditions including type 2 diabetes, heart disease, obstructive sleep apnea and certain cancers.

Surgery results in greater improvement in weight loss outcomes and obesity-related co-morbidities when compared with non-surgical interventions, regardless of the type of surgical procedure used. The most impressive change in bariatric procedure is the advent of laparoscopic sleeve gastrectomy (LSG). Since 2014, LSG has become the leading bariatric procedure in the USA.

Sleeve gastrectomy with loop bipartition ( SG+LB) was derived from the combined concepts of sleeve gastrectomy with transit bipartition (SG+TB), single anastomosis duodenal-ileostomy (SADI), mini-gastric bypass (MGB) and duodenal-jejunal bypass (DJB) with less nutritional and surgical complications.

Transit bipartition with sleeve gastrectomy (TB-SG) has been getting increased acceptance due to the advantage of preservation of the normal physiology and anatomy of duodenum. In iloe-duodenal sleeve bypass ,patients have a bypassed duodenum which is important in eliminating the foregut's negative incretin effects on insulin; however, this prevents any biliary access, if required later. TB-SG overcomes this problem by preserving the normal duodenal access, which makes the procedure more physiologic and easier to perform. With time, the gastroileal anastomosis has a tendency to enlarge resulting in "functional bypass" of duodenum, enhancing the anti-diabetic effect of the procedure.

* FIRSTLY,Sleeve gastrectomy technique:

  1. Positioning:

     It should be ensured that the operating table has the capacity to support the weight of the patient. The patient may be positioned supine or in French position with legs apart. The feet are secured to the foot board so that reverse trendelenburg position is possible. The arms should be well padded to prevent neurological injury should the arms be stretched out and secured to an arm board. Once the patient is strapped down, the table should be tilted to extremes to ensure that the patient is well secured and would not slip off the table.
  2. Decompression of the stomach:

     This can be achieved by insertion of orogastric tube, a hollow calibration tube by gastroscopy. The operators insert disposable 38 french calibration tube after positioning the patient and prior to draping. In doing so, surgeons are able to empty the gastric contents prior to surgery and during surgery, to maneuver the calibration tube to size the sleeve.
  3. Port placement:

     5 ports are typically inserted for LSG in our patients. A 10-12 optical trocar is inserted 20 cm below the left costal margin along the mid-clavicular line to gain access to the abdominal cavity. Other techniques like the use of Veress needle and open Hasson technique may be used. A 5mm epigastric port is inserted for introduction of a liver retractor. For patients where the distance between the xyphoid and umbilicus is up to 35cm we insert an infra-umbilical 15mm port as the working port for the surgeon. If the distance is more or the patient has central obesity this port is changed to a 10-12mm port that is placed approximately 20cm from xyphoid to the left of the mid line. Two 5mm ports are inserted in the left and right hypochondrial regions of the patient for assistant and surgeon.
  4. Measurement of the Antral pouch:

     Once pneumoperitoneum is established, a diagnostic laparoscopy is performed and hepatic steatosis assessed. The greater gastrocolic omentum is divided 5 cm from the pylorus with the aid of an energy device. There is consensus among bariatric surgeons that the antral pouch should be measured 2-6cm from the pylorus along greater curve as risk benefit ratio is best within these limits. However, some surgeons also believe that cutting too close to pylorus increases risk of leak and most would prefer to stay 4-6cm away.
  5. Devascularization:

     In the lateral technique, the devascularization process is continued up the greater curve of the stomach to the short gastric vessels with the help of the assistant who maintains traction and exposure during this process. Eventually, one reaches the left crus which is an important landmark of dissection. The left crus muscle is then routinely dissected and hiatus explored by some for a hernia, while others may differ. Surgeons selectively explore the hiatus of the symptomatic and endoscopically proven hiatus hernia as all our patients are evaluated for symptoms of reflux by questionnaire pre-operative and also have a gastroscopy performed. In patients with hiatus hernia, the hernia should be reduced and the defect repaired.

     In the medial approach, once the lesser sac is entered the process of stapling starts and devascularization is done only upon completion of sleeve.
  6. Gastric tube calibration:

     The 38 French Bougie inserted preoperatively is then advanced into the stomach along the lesser curve. This serves as the border of transection with the linear staple with the remnant lesser curve forming the neo- gastric pouch. One of the controversies lies in the optimal size of bougie to be used to size the sleeve.
  7. Creating the gastric tube:

     Linear transaction of the stomach can be performed using 3.5mm, 3.8 mm or 4.1 mm staples height depending on the thickness of the stomach wall. Any serosal tears during stapling or excessive unexpected bleeding should be carefully evaluated as it may be signaling a poorly stapled area.

     The use of staple-line reinforcement either through suturing or buttressing with biological or synthetic material is a hotly debated topic.
  8. Closure:

     The specimen is then delivered via the umbilical port. The staple line is then checked for any leaks; we do not routinely oversew the staple line. The 15mm port site is then closed with absorbable suture and the overlying skin stitched with a monofilament absorbable suture after local anesthesia is administered.
* SECONDLY,Combined sleeve gastrectomy and loop bipartition technique:

Sleeve gastrectomy is performed first, then a loop gastro-ileostomy 250-300 cm from the ileocecal valve or 200-250 cm from duodeno-jejunal junction was created at the dependent part of the antrum with 2 layers of handsewn suture but without division of the 1st part of duodenum. The resultant stomach tube has two outlets, one to the first part of duodenum through the pylorus and one to the terminal ileum through the gastroileostomy. The staple line and anastomosis was tested with methylene blue test at the end of the procedure.

Post-operative evaluation:

The patients will be followed up for a period for one year using the the same parameters as preoperative and the outcomes of each procedure will be collected and compared with each other ;

1. Regular follow up of weight and estimation of Excess Weight Loss (EWL).
2. Regular follow up of blood pressure.
3. Regular follow up of blood glucose and HbA1c.
4. Follow up investigations as serum electrolytes , iron studies and lipid profile.
5. Regular hospital follow up and strict adherence to nutritional supplementation and dietary instructions.
6. Follow up of outcomes for a period of one year; including effect on weight loss, and the resulting complications of each procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose body mass index (BMI) exceeds 40.
2. Patients with BMIs between 35 and 40 with high-risk co-morbid conditions or lifestyle-limiting obesity-induced physical conditions.
3. Age between 18 and 60 years old.
4. Both sexes.

Exclusion Criteria:

1. Patients younger than 18 and older than 60 years old.
2. BMI < 35.
3. Obesity due to medical diseases as hypothyroidism, cushing's , ……etc.
4. Surgically-unfit patients as those with contraindications to general anesthesia or uncorrectable coagulopathy.
5. Patients with limited life expectancy due to irreversible cardiopulmonary or other end-organ failure or metastatic or in-operable malignancy.
6. Patients who are pregnant or who expect to be pregnant within 12 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Comparison between sleeve gastrectomy and combined sleeve gastrectomy with loop bipartition (short-term outcomes). | one year
  Analysis of the effects of both stand-alone sleeve gastrectomy procedure and combined sleeve gastrectomy with loop bipartition on weight loss and obesity-related hypertension and diabetes mellitus, and also the complications associated with each procedure .

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt